CLINICAL TRIAL: NCT01515865
Title: A Phase 4, Randomized-withdrawal, Double-blind, Placebo Controlled, Parallel-group Study to Investigate the Clinical Benefit of Midodrine Hydrochloride in Male and Female Subjects With Symptomatic Orthostatic Hypotension
Brief Title: Clinical Efficacy of Midodrine in Symptomatic Orthostatic Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD426-405; 2012-005760-99 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Symptomatic Orthostatic Hypotension
MeSH Terms: interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midodrine HCl (Experimental)
  Interventions: Drug: Midodrine HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine HCl — dose at subject's current dose level
  Other Names: ProAmatine®
  Arms: Midodrine HCl
Drug: Placebo — single dose of matching placebo
  Arms: Placebo

SUMMARY:
To study the effect of midodrine against the symptoms of orthostatic hypotension

DETAILED DESCRIPTION:
The efficacy of midodrine will be assessed in those subjects who have severe symptoms of orthostatic hypotension when not taking midodrine and are controlled when taking midodrine. The study will involve approximately 9 overnight stays.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects must be 18 years of age or older and ambulatory.
2. Females of child-bearing potential (FOCP) must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test.
3. A documented history of severe Symptomatic Orthostatic Hypotension (SOH) that, in the judgment of the treating physician, has required treatment with midodrine HCl, and has been at a stable dose for at least 3 months.
4. The subject has manifested at least 1 of the following symptoms while standing or had a medical history of 1 of the following when not treated for orthostatic hypotension (OH): dizziness, lightheadedness, feeling faint, or feeling like they might black out.

Exclusion criteria

1. The subject is a pregnant or lactating female.
2. The subject has pre-existing sustained supine hypertension greater than 180mmHg systolic and 110mmHg diastolic BP or had these measurements at the Screening Visit. Sustained is defined as persistently greater at 2 separate measurements at least 5 minutes apart with the subject supine and at rest for the 5 minutes.
3. Subjects taking concomitant medications of interest are excluded unless those medications are reviewed and discussed with the Medical Monitor or Study Physician and documented prior to enrolling the subject. If agreement is reached between the Investigator and Sponsor for the subject to continue in the study, all allowed medications should be maintained at a constant dose throughout the study.
4. The Principal Investigator deems any clinical laboratory test (at the Screening Visit) abnormality to be clinically significant
5. The subject has participated in other studies of investigational drugs or devices within 30 days prior to enrollment in this study (other than Study SPD426-406).
6. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
7. The subject has a concurrent chronic or acute illness, disability, or other condition (including significant unexpected laboratory or electrocardiogram [ECG] findings) that might confound the results of the tests and/or measurements administered in this study, or that might have increased the risk to the subject.
8. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
9. Prior enrollment failure or randomization in this study.
10. History of alcohol abuse or other substance abuse within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2013-11-11 (Actual); Study Completion 2013-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- United States (18):
  - California Clinical Trials Medical Group, Glendale, California
  - Pharmaseek-Burbank, North Hollywood, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Advance Research Institute Inc, New Port Richey, Florida
  - DMI Reasearch Inc, Pinellas Park, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Chicago Medical VA, North Chicago, Illinois
  - Analab Clinical Research Inc, Lenexa, Kansas
  - PAREXEL International - Baltimore EPCU Harbor Hospital, Baltimore, Maryland
  - Frontage Clinical Services, Hackensack, New Jersey
  - Buffalo Clinical Research Center (BCRC), Buffalo, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Kidney and Hypertension Center, Roseburg, Oregon
  - New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee
  - UT South West Medical Center, Dallas, Texas
  - The Heartbeat Clinic, PA, McKinney, Texas
  - Aspen Clinical Research, Orem, Utah
- Czechia (3):
  - Fakultní nemocnice Hradec Králové, Hradec, Králové
  - Fakultní nemocnice Ostrava, Ostrava, Poruba
  - Fakultní nemocnice v Motole, Prague
- Poland (5):
  - EMC Silesia Sp. z o.o.; NZOZ Szpital Geriatryczny im. Jana Pawła II w Katowicach, Katowice
  - Specjalistyczna Praktyka Lekarska Prof. Grzegorz Opala, + satelite site:NZOZ Szpital Avimed Sp. z o.o., Katowice
  - Centrum Medyczne HCP, Lecznictwo Stacjonarne, Oddział Udarowy, Poznan
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Wojskowy Instytut Medyczny, Klinika Neurologiczna, Warsaw
- Slovakia (6):
  - Neurologická klinika SZU a UNB, Univerzitná nemocnica Bratislava, Bratislava
  - Neurologická klinika UN Martin, Univerzitná nemocnica Martin, Martin
  - Neurologická klinika FN Nitra, Fakultná nemocnica Nitra, Nitra
  - Neurologické oddelenie, Nemocnica s poliklinikou Spišská Nová Ves, a.s., Spišská Nová Ves
  - Neurologické oddelenie FN Trnava, Fakultná nemocnica Trnava, Trnava
  - Neurologické oddelenie FNsP Žilina, Fakultná nemocnica s poliklinikou Žilina, Žilina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received the dose and frequency of Midodrine HCl that they had been receiving during their non-study treatment prior to enrolling in this study.
Groups:
- Midodrine HCl - (Open-label): On the morning of Day -1, subjects took their usual morning dose of midodrine HCl, using their own midodrine HCl supplies at approximately the same time before rising that they would normally take their morning dose. On the morning of Day 1, subjects had their usual morning dose of midodrine HCl withheld. On Day 2, all eligible subjects continued on their midodrine HCl dose regimen over at least 14 days, using study-supplied investigational product.
- Midodrine HCl - (Randomized): On Day 16 subjects received over-encapsulated midodrine HCl tablets (equivalent to their previously prescribed dose).
- Placebo - (Randomized): On Day 16 subjects received matching placebo.
Period: Part A (Open-label)
Arm/Group | Midodrine HCl - (Open-label) | Midodrine HCl - (Randomized) | Placebo - (Randomized)
Started | 98 | 0 | 0
Completed | 95 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Other | 3 | 0 | 0
Period: Part B (Open-label)
Arm/Group | Midodrine HCl - (Open-label) | Midodrine HCl - (Randomized) | Placebo - (Randomized)
Started | 71 (Twenty-four subjects from Part A did not meet the criteria required to be enrolled into Part B.) | 0 | 0
Completed | 69 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Part C (Randomized)
Arm/Group | Midodrine HCl - (Open-label) | Midodrine HCl - (Randomized) | Placebo - (Randomized)
Started | 0 | 33 (A total of two subjects from Part B did not meet the criteria required to be enrolled into Part C.) | 34
Completed | 0 | 33 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Enrolled Population consisted of all subjects who participated in Part A baseline procedures starting at Day -1.
Arm/Group | Enrolled Population
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (17.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90
  Slovakia | 3
  Poland | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Failed to Maintain a Response
Description: Failure to maintain a response was defined as any randomized subject that met both criterion 1 and criterion 2 below on Day 16: 1. The Orthostatic Hypotension Symptom Assessment (OHSA) Item 1 score increased by >=4 points compared to baseline. OHSA Item 1 is a dizziness scale that is scored on a range from 0 (no dizziness) to 10 (severe dizziness). A lower score indicates less severe symptoms. 2. There was an increase in the number of syncopal/near syncopal events or severity of events within 15 minutes of standing compared to those observed at baseline. Syncope was defined as a loss of consciousness, and near syncope was defined as a feeling (e.g., dizziness, lightheadedness, feeling faint, feeling as though one would black out) that, without intervention, would lead to a loss of consciousness.
Time Frame: 30 minutes post-dose on Day 16
Population: The Full Analysis Set was defined as all randomized subjects who received at least 1 dose of double-blind investigational product.
Measure: Number; unit: percentage of participants
Groups:
- Midodrine HCl: Over-encapsulated midodrine HCl tablet at the subjects previously prescribed dose level.
- Placebo: Matching placebo treatment (utilizing the same number of placebo capsules that would be required to constitute their midodrine HCl dose).
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 33 | 34
percentage of participants | 30.3 | 44.1
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.3145, Fisher Exact; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-37.6 to 9.8]

ADVERSE EVENTS:
Groups:
- Midodrine HCl - Open-label (Part A): dose at the subjects current dose level
- Midodrine HCl - Open-label (Part B): open-label study-supplied (Part B) dose at subjects current dose level
- Midodrine HCl - Randomized (Part C): over-encapsulated randomized dose (Part C) at subjects current dose level
- Placebo - Randomized (Part C): over-encapsulated randomized matching placebo
Arm/Group | Midodrine HCl - Open-label (Part A) | Midodrine HCl - Open-label (Part B) | Midodrine HCl - Randomized (Part C) | Placebo - Randomized (Part C)
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/71 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 5/98 | 2/71 | 0/33 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine HCl - Open-label (Part A) (N=98) | Midodrine HCl - Open-label (Part B) (N=71) | Midodrine HCl - Randomized (Part C) (N=33) | Placebo - Randomized (Part C) (N=34)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.